CLINICAL TRIAL: NCT06269237
Title: Point of Care Test of LTA Level in Tear Fluid, Measured With a POCT Test, in DE Patients Following IPL Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023LTA
Record Dates: First submitted 2023-06-03; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-05

CONDITIONS: Dry Eye
Keywords: dry eye; intense pulsed light; Lymphotoxin alpha
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPL (Experimental): Participants in the group with 3 sessions of IPL, 2 weeks apart.
  Interventions: Device: M22
- control (Sham Comparator): Participants in the group with 2 sessions of IPL, 1 session of sham IPL, 2 weeks apart.
  Interventions: Device: M22; Device: sham M22

INTERVENTIONS:
Device: M22 — Participants in the group with 3 sessions of IPL, 2 weeks apart. Device: Intense pulsed light IPL treatment intensity was chosen based on the Fitzpatrick scale as follows: Fitzpatrick scale I, II, III, 10-15 J/cm2 with a 570-nm filter.
  Other Names:
  • IPL
Device: sham M22 — Participants in the group with 2 sessions of IPL, 1 session of sham IPL, 2 weeks apart. Device: Intense pulsed light IPL treatment intensity was chosen based on the Fitzpatrick scale as follows: Fitzpatrick scale I, II, III, 10-15 J/cm2 with a 570-nm filter.
  Arms: control

SUMMARY:
To quantify and compare tear levels of Intense pulsed light (IPL) and traditional dry eye clinical tests in dry eye patients before and after Intense pulsed light (IPL) treatment.

DETAILED DESCRIPTION:
Dry eye is multifactorial, mainly manifested as eye pain, visual impairment (blurred and blurry vision), tear film instability, and tear film hypertonicity, which can cause ocular surface damage. Some possible causes of DED include aging, menopause, Meibomian gland dysfunction (Meibomian gland dysfunction; MGD), Sjogren's syndrome, conjunctival fibrotic disease, refractive surgery, and systemic or topical drugs. Insufficient tear secretion or excessive tear evaporation has been demonstrated to cause precorneal tear concentration or hypertonicity, which disrupts tear film homeostasis. Tear film hypertonicity can cause cell morphological changes, inflammatory cascades, cell death, tear film instability, and further lead to tear hypertonicity. Mgd-induced Evaporative dry eye; EDE) is the most common form of dry eye]. Anti-inflammatory drugs, antibiotics, hot compress, eyelid cleaning and meibomian gland expression are the treatment standards for MGD. However, its long-term efficacy is not satisfactory due to poor patient compliance.

MGD has been found to be associated with eyelid inflammatory disorders. Rosacea affects 5.46% of adults (range 0.09-24.1%) of whom 58% have MGD. Ocular symptoms precede cutaneous rosacea in 15 to 10% of cases, indicating the presence of subclinical variation.

Intense pulsed light (IPL) has mostly been utilized as a dermatological treatment for conditions like facial rosacea, facial erythema, acne, and seborrheic keratosis throughout the last few decades. In 2015, researchers reported the use of IPL for treating MGD to improve the signs and symptoms of DED. Two years later, the TFOS DEWS II report listed IPL as an option for treating DED. Mechanisms of IPL action include liquefication of meibum, regulate inflammation, destroy abnormal blood vessels, inhibit metalloproteinases, and photo modulation. Past studies have reported that IPL treatment modulates tear inflammatory cytokines, with improvements in tear inflammation prior to changes in dry eye signs, however, these studies have been limited by laboratory tests. It is difficult to apply in clinical practice.

Lymphotoxin-alpha (LTA) is a member of the tumor necrosis factor (TNF) superfamily and is expressed by a variety of cells, including T cells, B cells and natural killer cells. LTA secreted to the extracellular space assembles into a homotrimer (LTα3) as a soluble protein, and binds to the tumor necrosis factor receptor to play a role. LTA has been shown to be a diagnostic biomarker for dry eye in past studies. The aim of this study is to investigate the therapeutic mechanism of IPL and provide evidence for the treatment of dry eye by using a point-of-care LTA detection reagent to quantitatively compare the tear LTA levels before and after IPL treatment with traditional dry eye clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* Fitzpatrick skin types I to IV
* capable and willing to comply with the treatment and follow-up obligations
* a determination of DED based on (a) the Ocular Surface Disease Index (OSDI) ≥13 score represents severe DED, (b) non-invasive tear film breakup time (NITBUT) of ≤5 sec, or conjunctivocorneal staining score (CS) ≥3 points according to the Japanese Dry Eye Consensus

Exclusion Criteria:

* Existing ocular trauma, infectious diseases, recent surgical history
* Skin defects, pigmentation, moles, scars in the treatment area, skin cancer
* Autoimmune diseases, skin allergies.
* Pregnancy or lactation
* Fitzpatrick skin type V or VI.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-22 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
LTA | Day-0 (baseline), day-21, day-42, day-63 and day-84
  Lymphotoxin-alpha (LTA) is a member of the tumor necrosisfactor (TNF) superfamily and is expressed by a variety of cells, including T cells, B cells and natural killer cells. LTA secreted to the extracellular space assembles into a homotrimer (LTα3) as a soluble protein [23], and binds to the tumor necrosis factor receptor to play a role. LTA will be measured using an immunochromatography assay by collecting 1ul tear samples from the lateral canthus using a capillary tear collector. To assess the concentration of LTA in the tear samples, a commercial reagent card (S05B, Seinda Biomedical Corporation, Guangdong, China) based on colloidal gold and immunochromatographic analysis was utilized.
Non-invasive tear break-up time (NITBUT) | Day-0 (baseline), day-21, day-42, day-63 and day-84
  Non-invasive initial tear film breaking time will be assessed using the Keratograph 5M (Oculus, Germany) topographer.
  Three sequentially readings will be captured, and the median value will be included in the final analysis. The median value will be recorded.

SECONDARY OUTCOMES:
Fluorescein and lissamine conjunctival and cornea staining (CFS) | Day-0 (baseline), day-21, day-42, day-63 and day-84
  Fluorescein and lissamine staining of the ocular surface will be divided into three zones comprising nasal conjunctival, corneal, and temporal conjunctival areas. The staining score ranged from 0 to 3 for each zone, yielding a total score of 0-9 for the ocular surface. Higher scores means worse.
Meibomian quality | Day-0 (baseline), day-21, day-42, day-63 and day-84
  Meibum quality will be assessed under a slit-lamp: Five meibomian gland in the middle parts of the eyelid will be assessed using a scale of 0 to 3 for each gland (0 represented clear meibum; 1 represented cloudy meibum; 2 represented cloudy and granular meibum; and 3 represented thick, toothpaste like consistency meibum)
Tear Film Lipid Layer Score(TFLL) | Day-0 (baseline), day-21, day-42, day-63 and day-84
  Tear Film Lipid Layer interferometry will be assessed using DR-1 (Kowa, Nagoya, Japan). The results will be graded as follows: grade 1, somewhat gray color, uniform distribution; grade 2, somewhat gray color, nonuniform distribution; grade 3, a few colors, nonuniform distribution; grade 4, many colors, nonuniform distribution; grade 5, corneal surface partially exposed.
Tear meniscus height (TMH) | Day-0 (baseline), day-21, day-42, day-63 and day-84
  TMH using the Keratograph 5M (Oculus, Germany) topographer will be measured three times consecutively and the median value was recorded.
Conjunctival hyperemia (RS score) | Day-0 (baseline), day-21, day-42, day-63 and day-84
  Conjunctival hyperemia (RS score) will be assessed by Keratograph image (Oculus, Germany) of 1156*873 pixels, redness score (RS) (accurate to 0.1 U) was displayed on the computer screen that ranged from 0.0 (normal) to 4.0 (severe).
Ocular Surface Disease Index (OSDI) | Day-0 (baseline), day-21, day-42, day-63 and day-84
  The patient will answer each question on a scale ranging from 0 to 4, with 0 indicating 'none of the time' and 4 indicating 'all of the time'. If a certain question is deemed irrelevant, it will be marked as 'not applicable (N/A)' and excluded from the analysis. The OSDI total score is calculated according to the following formula. The scale ranges from 0 to 100, with higher scores representing more severe cases of dry eye syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Guanghao Qin, Study Chair — He Eye Hospital

IPD SHARING:
Plan to Share IPD: Yes
The study's findings will be shared regardless of the effect's direction. All possible beneficiaries of the research, including patients, carers, family, doctors, advisory boards, and medical boards, will receive trial data. Publications in high impact, open-access medical journals and talks at national and international medical conferences will serve this purpose.
Supporting Information: Study Protocol, SAP
Time Frame: The Steering Committee will write and submit the report for publication at the end of the study
Access Criteria: Use in clinical studies

REFERENCES:
- [Background] Tsubota K, Yokoi N, Shimazaki J, Watanabe H, Dogru M, Yamada M, Kinoshita S, Kim HM, Tchah HW, Hyon JY, Yoon KC, Seo KY, Sun X, Chen W, Liang L, Li M, Liu Z; Asia Dry Eye Society. New Perspectives on Dry Eye Definition and Diagnosis: A Consensus Report by the Asia Dry Eye Society. Ocul Surf. 2017 Jan;15(1):65-76. doi: 10.1016/j.jtos.2016.09.003. Epub 2016 Oct 8. PMID 27725302
- [Background] Schein OD, Munoz B, Tielsch JM, Bandeen-Roche K, West S. Prevalence of dry eye among the elderly. Am J Ophthalmol. 1997 Dec;124(6):723-8. doi: 10.1016/s0002-9394(14)71688-5. PMID 9402817
- [Background] Evans V, Millar TJ, Eden JA, Willcox MD. Menopause, hormone replacement therapy and tear function. Adv Exp Med Biol. 2002;506(Pt B):1029-33. doi: 10.1007/978-1-4615-0717-8_145. No abstract available. PMID 12614027
- [Background] Valencia-Nieto L, Novo-Diez A, Blanco-Vazquez M, Lopez-Miguel A. Therapeutic Instruments Targeting Meibomian Gland Dysfunction. Ophthalmol Ther. 2020 Dec;9(4):797-807. doi: 10.1007/s40123-020-00304-3. Epub 2020 Sep 24. PMID 32968960
- [Background] Kang YS, Lee HS, Li Y, Choi W, Yoon KC. Manifestation of meibomian gland dysfunction in patients with Sjogren's syndrome, non-Sjogren's dry eye, and non-dry eye controls. Int Ophthalmol. 2018 Jun;38(3):1161-1167. doi: 10.1007/s10792-017-0577-4. Epub 2017 May 31. PMID 28567496
- [Background] Sambhi RS, Sambhi GDS, Mather R, Malvankar-Mehta MS. Dry eye after refractive surgery: a meta-analysis. Can J Ophthalmol. 2020 Apr;55(2):99-106. doi: 10.1016/j.jcjo.2019.07.005. Epub 2019 Aug 20. PMID 31712000
- [Background] Fraunfelder FT, Sciubba JJ, Mathers WD. The role of medications in causing dry eye. J Ophthalmol. 2012;2012:285851. doi: 10.1155/2012/285851. Epub 2012 Aug 27. PMID 23050121
- [Background] Askeroglu U, Alleyne B, Guyuron B. Pharmaceutical and herbal products that may contribute to dry eyes. Plast Reconstr Surg. 2013 Jan;131(1):159-167. doi: 10.1097/PRS.0b013e318272a00e. PMID 23271525
- [Background] Bron AJ, de Paiva CS, Chauhan SK, Bonini S, Gabison EE, Jain S, Knop E, Markoulli M, Ogawa Y, Perez V, Uchino Y, Yokoi N, Zoukhri D, Sullivan DA. TFOS DEWS II pathophysiology report. Ocul Surf. 2017 Jul;15(3):438-510. doi: 10.1016/j.jtos.2017.05.011. Epub 2017 Jul 20. PMID 28736340
- [Background] Thode AR, Latkany RA. Current and Emerging Therapeutic Strategies for the Treatment of Meibomian Gland Dysfunction (MGD). Drugs. 2015 Jul;75(11):1177-85. doi: 10.1007/s40265-015-0432-8. PMID 26130187
- [Background] Machalinska A, Zakrzewska A, Markowska A, Safranow K, Wiszniewska B, Parafiniuk M, Machalinski B. Morphological and Functional Evaluation of Meibomian Gland Dysfunction in Rosacea Patients. Curr Eye Res. 2016 Aug;41(8):1029-1034. doi: 10.3109/02713683.2015.1088953. Epub 2015 Dec 7. PMID 26644191
- [Background] Tavassoli S, Wong N, Chan E. Ocular manifestations of rosacea: A clinical review. Clin Exp Ophthalmol. 2021 Mar;49(2):104-117. doi: 10.1111/ceo.13900. Epub 2021 Feb 3. PMID 33403718
- [Background] Viso E, Rodriguez-Ares MT, Abelenda D, Oubina B, Gude F. Prevalence of asymptomatic and symptomatic meibomian gland dysfunction in the general population of Spain. Invest Ophthalmol Vis Sci. 2012 May 4;53(6):2601-6. doi: 10.1167/iovs.11-9228. PMID 22427596
- [Background] Yang L, Pazo EE, Zhang Q, Wu Y, Song Y, Qin G, Zhang H, Li J, Xu L, He W. Treatment of contact lens related dry eye with intense pulsed light. Cont Lens Anterior Eye. 2022 Apr;45(2):101449. doi: 10.1016/j.clae.2021.101449. Epub 2021 Apr 28. PMID 33933353
- [Background] Rong B, Tang Y, Liu R, Tu P, Qiao J, Song W, Yan X. Long-Term Effects of Intense Pulsed Light Combined with Meibomian Gland Expression in the Treatment of Meibomian Gland Dysfunction. Photomed Laser Surg. 2018 Oct;36(10):562-567. doi: 10.1089/pho.2018.4499. Epub 2018 Sep 22. PMID 30251914
- [Background] Dell SJ, Gaster RN, Barbarino SC, Cunningham DN. Prospective evaluation of intense pulsed light and meibomian gland expression efficacy on relieving signs and symptoms of dry eye disease due to meibomian gland dysfunction. Clin Ophthalmol. 2017 May 2;11:817-827. doi: 10.2147/OPTH.S130706. eCollection 2017. PMID 28496300
- [Background] Weiss RA, Ross EV, Tanghetti EA, Vasily DB, Childs JJ, Smirnov MZ, Altshuler GB. Characterization of an optimized light source and comparison to pulsed dye laser for superficial and deep vessel clearance. Lasers Surg Med. 2011 Feb;43(2):92-8. doi: 10.1002/lsm.21032. PMID 21384389
- [Background] Taudorf EH, Olsen J, Lindso Andersen P, Bouazzi D, Jemec GBE. Dynamic Optical Coherence Tomography Imaging of Telangiectasia Prior to Intense Pulsed Light Treatment-An Opportunity to Target Treatment? Lasers Surg Med. 2021 Feb;53(2):212-218. doi: 10.1002/lsm.23280. Epub 2020 Jun 12. PMID 32533557
- [Background] Wang B, Wu Y, Luo YJ, Xu XG, Xu TH, Chen JZ, Gao XH, Chen HD, Li YH. Combination of intense pulsed light and fractional CO(2) laser treatments for patients with acne with inflammatory and scarring lesions. Clin Exp Dermatol. 2013 Jun;38(4):344-51. doi: 10.1111/ced.12010. Epub 2013 Apr 3. PMID 23551214
- [Background] Liu R, Rong B, Tu P, Tang Y, Song W, Toyos R, Toyos M, Yan X. Analysis of Cytokine Levels in Tears and Clinical Correlations After Intense Pulsed Light Treating Meibomian Gland Dysfunction. Am J Ophthalmol. 2017 Nov;183:81-90. doi: 10.1016/j.ajo.2017.08.021. Epub 2017 Sep 6. PMID 28887117
- [Background] Liu J, Liu L, Zhou L, Chen L, Chen X, Xiong X, Deng Y. The Effect of Intense Pulsed Light on the Skin Microbiota and Epidermal Barrier in Patients with Mild to Moderate Acne Vulgaris. Lasers Surg Med. 2021 Dec;53(10):1348-1355. doi: 10.1002/lsm.23426. Epub 2021 Jul 5. PMID 34224604
- [Background] Li Q, Liu J, Liu C, Piao J, Yang W, An N, Zhu J. Effects of intense pulsed light treatment on tear cytokines and clinical outcomes in meibomian gland dysfunction. PLoS One. 2021 Aug 26;16(8):e0256533. doi: 10.1371/journal.pone.0256533. eCollection 2021. PMID 34437596
- [Background] Chen H, Chen H, Liang L, Zhong Y, Liang Y, Yu Y, Huang S, Lu X. Evaluation of Tear Protein Markers in Dry Eye Disease with Different Lymphotoxin-Alpha Expression Levels. Am J Ophthalmol. 2020 Sep;217:198-211. doi: 10.1016/j.ajo.2020.03.013. Epub 2020 Mar 21. PMID 32209340
- [Background] Uchino Y, Uchino M, Dogru M, Ward S, Yokoi N, Tsubota K. Changes in dry eye diagnostic status following implementation of revised Japanese dry eye diagnostic criteria. Jpn J Ophthalmol. 2012 Jan;56(1):8-13. doi: 10.1007/s10384-011-0099-y. Epub 2011 Nov 15. PMID 22080359
- [Background] Arita R, Itoh K, Inoue K, Amano S. Noncontact infrared meibography to document age-related changes of the meibomian glands in a normal population. Ophthalmology. 2008 May;115(5):911-5. doi: 10.1016/j.ophtha.2007.06.031. PMID 18452765
- [Background] Yokoi N, Takehisa Y, Kinoshita S. Correlation of tear lipid layer interference patterns with the diagnosis and severity of dry eye. Am J Ophthalmol. 1996 Dec;122(6):818-24. doi: 10.1016/s0002-9394(14)70378-2. PMID 8956636
- [Background] Ma J, Li C, Zhao Y, Shen Z, Hu B, Peng R, Hong J. Ophthalmic manifestations are associated with reduced tear lymphotoxin-alpha levels in chronic ocular graft-versus-host disease. BMC Ophthalmol. 2022 Jan 10;22(1):18. doi: 10.1186/s12886-022-02251-y. PMID 35012541
- [Background] Chen X, Graham J, Dabbah MA, Petropoulos IN, Tavakoli M, Malik RA. An Automatic Tool for Quantification of Nerve Fibers in Corneal Confocal Microscopy Images. IEEE Trans Biomed Eng. 2017 Apr;64(4):786-794. doi: 10.1109/TBME.2016.2573642. Epub 2016 Jun 7. PMID 27295646
- [Background] Zhang XM, Yang LT, Zhang Q, Fan QX, Zhang C, You Y, Zhang CG, Lin TZ, Xu L, Moutari S, Moore JE, Pazo EE, He W. Reliability of Chinese web-based ocular surface disease index questionnaire in dry eye patients: a randomized, crossover study. Int J Ophthalmol. 2021 Jun 18;14(6):834-843. doi: 10.18240/ijo.2021.06.07. eCollection 2021. PMID 34150537